CLINICAL TRIAL: NCT06383390
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Event-Driven Study to Investigate the Effect of Retatrutide on the Incidence of Major Adverse Cardiovascular Events and Major Adverse Kidney Events in Participants With Body Mass Index ≥27 kg/m2 and Atherosclerotic Cardiovascular Disease and/or Chronic Kidney Disease
Brief Title: The Effect of Retatrutide Once Weekly on Cardiovascular Outcomes and Kidney Outcomes in Adults Living With Obesity (TRIUMPH-Outcomes)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18584; J1I-MC-GZBO (Other: Eli Lilly and Company); 2023-508630-34-00 (Other: EU CTR Number)
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Atherosclerotic Cardiovascular Disease (ASCVD); Chronic Kidney Disease (CKD)
Keywords: Cardiovascular Disease; Kidney Disease; Major Adverse Cardiovascular Events (MACE); Renal Outcomes; Cardiovascular Risk Reduction; Kidney Disease Progression; Cardiometabolic Risk Factors; Cardiovascular Outcomes; Kidney Outcomes; Type 2 Diabetes; Heart Disease; Coronary Artery Disease; Cerebrovascular Disease; Peripheral Arterial Disease; Nonfatal Myocardial Infarction (MI); Nonfatal Stroke; Cardiovascular (CV) Death; Hospitalization or Urgent Visit Due to Heart Failure (HF); Renal Death; End Stage Kidney Disease (ESKD)
MeSH Terms: conditions — Atherosclerosis; Renal Insufficiency, Chronic; Cardiovascular Diseases; Kidney Diseases; Diabetes Mellitus, Type 2; Heart Diseases; Coronary Artery Disease; Cerebrovascular Disorders; Peripheral Arterial Disease; Death; Kidney Failure, Chronic | interventions — retatrutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Retatrutide (Experimental): Participants will receive escalated doses of retatrutide administered subcutaneously (SC) up to a maximum tolerated dose.
  Interventions: Drug: Retatrutide
- Placebo (Placebo Comparator): Participants will receive matching placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Retatrutide — Administered SC
  Other Names: LY3437943
  Arms: Retatrutide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine if retatrutide can significantly lower the incidence of serious heart-related complications or prevent the worsening of kidney function. The trial will enroll adults with body mass index 27 kg/m^2 or higher and Atherosclerotic Cardiovascular Disease and/or chronic kidney disease. The study will last for about 5 years. Participants will have up to 27 clinic visits with the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Participants may be without type 2 diabetes (T2D), or with T2D if their hemoglobin A1c (HbA1c) is 10% or lower
* Participants have established atherosclerotic cardiovascular disease (ASCVD) and/or chronic kidney disease (CKD), as evidenced at least one of the following:

  * Coronary artery disease
  * Cerebrovascular disease
  * Peripheral arterial disease
  * Chronic kidney disease defined as:

    * eGFR <45 millilitres/minute/1.73 meter squared (mL/min/1.73m^2) and UACR >30 milligram/gram (mg/g) (0.030 mg/mg)
    * eGFR <60 mL/min/1.73 m^2 and UACR >100 mg/g (0.100 mg/mg), or
    * eGFR <75 mL/min/1.73 m^2 and UACR >300 mg/g (0.300 mg/mg) (eGFR is calculated by central lab based on Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine-cystatin c equation as determined by central lab)
* A Body Mass Index of ≥27.0 kilograms per meter squared (kg/m^2)

Exclusion Criteria:

Diabetes related:

* Participants have Type 1 Diabetes or any history of diabetic ketoacidosis

CV related:

* Participants have any of the following cardiovascular conditions ≤ 90 days prior to randomization:

  * Myocardial infarction
  * Acute coronary syndrome
  * Stroke, or
  * Coronary, peripheral, or carotid artery arterial revascularization procedure.
* Have acute decompensated heart failure requiring hospitalization.
* Have New York Heart Association (NYHA) Classification Class IV heart failure at screening

Kidney related:

* Participants have an eGFR <20 mL/min/1.73 m^2 at screening
* Have UACR >5000 mg/g (5.000 mg/mg) at screening
* Have received any form of dialysis ≤ 90 days from the date of randomization
* Have either undergone a kidney transplant or have a transplant procedure scheduled

Other medical conditions:

* Participants have had or plan to have a surgical treatment for obesity,
* Have a history of chronic or acute pancreatitis
* Have a family or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia (MEN) syndrome type 2
* Have a known clinically significant gastric emptying abnormality, such as severe gastroparesis or gastric outlet obstruction

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Time to First Occurrence of Composite Endpoints | Randomization up to Study Completion (Approximate 248 Weeks)
  A composite endpoint includes nonfatal myocardial infarction (MI), nonfatal stroke, cardiovascular (CV) death, or hospitalization or urgent visit due to heart failure (HF).
Time to First Occurrence of Composite Endpoint of End Stage Kidney Disease (ESKD), ≥ 40% Sustained Decline in Estimated Glomerular Filtration Rate (eGFR), CV Death or Renal Death | Randomization up to Study Completion (Approximate 248 Weeks)
  ESKD is defined as the following individual components: persistent eGFR <15 mL/min/1.73 m^2 confirmed by 2 measurements at least 4 weeks apart at the central laboratory, initiation of dialysis for at least 28 days, receiving a kidney transplant.
  Sustained decline in eGFR (≥40%) will be confirmed by a repeated measure at least 4 weeks after the first result.

SECONDARY OUTCOMES:
Time to First Occurrence of Composite Endpoint of Major Cardiovascular Events (MACE-3) | Randomization up to Study Completion (Approximate 248 Weeks)
  MACE-3 includes CV death, nonfatal MI, and nonfatal stroke.
Time to First Occurrence of Composite Endpoint of CV death, or hospitalization or urgent visit due to HF | Randomization up to Study Completion (Approximate 248 Weeks)
  Time to First Occurrence of Composite Endpoint of CV death, or hospitalization or urgent visit due to HF.
Time to Occurrence of All-Cause Death | Randomization up to Study Completion (Approximate 248 Weeks)
  Time to all-cause death.
Time to First Occurrence of composite endpoint of ≥ 40% Sustained Decline in eGFR, End-Stage Renal Disease (ESRD), or Renal Death | Randomization up to Study Completion (Approximate 248 Weeks)
Percentage change from Baseline in Albuminuria urinary albumin/creatinine ratio (UACR) in Participants with UACR ≥30 mg/g (0.03 mg/mg) at baseline | Randomization up to Study Completion (Approximate 248 Weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (741):
- United States (205):
  - Alabama Kidney Research, Alabaster, Alabama
  - Central Research Associates, Birmingham, Alabama
  - Alliance for Multispecialty Research, LLC, Daphne, Alabama
  - Nephrology Consultants, Huntsville, Alabama
  - Alliance for Multispecialty Research, LLC, Mobile, Alabama
  - Prime Medical Group, LLC dba Gilbert Center for Family Medicine, LLC, Gilbert, Arizona
  - Sun City Clinical Research, Glendale, Arizona
  - Arizona Kidney Disease & Hypertension Center (AKDHC) - Thunderbird, Glendale, Arizona
  - Helios Clinical Research - SAZ-PDV-026, Paradise Valley, Arizona
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - Phoenix Clinical LLC, Phoenix, Arizona
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Absolute Clinical Research, Phoenix, Arizona
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Clinical Research Institute of Arizona (CRI) - Sun City West, Sun City West, Arizona
  - Synexus Clinical Research US, Inc./Orange Grove Family Practice, Tucson, Arizona
  - Cardiology and Medicine Clinic, Little Rock, Arkansas
  - Kidney & Hypertension Center - Apple Valley, Apple Valley, California
  - Invivo - Bakersfield, Bakersfield, California
  - American Institute of Research, Beverly Hills, California
  - Hope Clinical Research, Inc., Canoga Park, California
  - Valley Clinical Trials, Inc., Covina, California
  - North Coast Cardiology, Encinitas, California
  - Neighborhood Healthcare Institute of Health, Escondido, California
  - HB Clinical Trials - Fountain Valley, Fountain Valley, California
  - Care Access - Huntington Beach, Huntington Beach, California
  - Irvine Clinical Research, Irvine, California
  - Scripps Whittier Diabetes Institute, La Jolla, California
  - Long Beach Research Institute, Long Beach, California
  - Ark Clinical Research, Long Beach, California
  - North America Research Institute, Lynwood, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Desert Oasis Healthcare Medical Group, Palm Springs, California
  - California Liver Research Institute, Pasadena, California
  - Western University of Health Sciences, Pomona, California
  - California Kidney Specialists, San Dimas, California
  - Southern California Clinical Research, Santa Ana, California
  - Care Access - Santa Clarita, Santa Clarita, California
  - Encompass Clinical Research, Spring Valley, California
  - Valiance Clinical Research, Tarzana, California
  - Care Access - Thousand Oaks, Thousand Oaks, California
  - Med Partners, Inc. dba Premiere Medical Center of Burbank, Inc., Toluca Lake, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - UCLA South Bay Endocrinology, Torrance, California
  - InvivoCure, Van Nuys, California
  - National Institute of Clinical Research (NICR) - High Desert, Victorville, California
  - Synexus Clinical Research US, Inc., Vista, California
  - Millennium Clinical Trials, Westlake Village, California
  - Western Nephrology, Arvada, Colorado
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Cardiology Associates of Fairfield County, P.C., Stamford, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - American Research Institute, Cutler Bay, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Jellinger and Lerman, MD PA dba The Center for Diabetes and Endocrine Care, Fort Lauderdale, Florida
  - Florida Kidney Physicians - Fort Lauderdale, Fort Lauderdale, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Lakeview Institute of Clinical Research, Leesburg, Florida
  - Flourish Research - Miami, LLC, Miami, Florida
  - New Age Medical Research Corporation, Miami, Florida
  - Onhealth Research Center, Miami, Florida
  - Inpatient Research Clinic, Miami Lakes, Florida
  - CTR Oakwater, LLC, Orlando, Florida
  - Omega Research Orlando, Orlando, Florida
  - Florida Kidney Physicians, LLC, Port Charlotte, Florida
  - Florida Kidney Physicians - Tampa, Riverview, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Care Access - Tamarac, Tamarac, Florida
  - MOORE Clinical Research, Inc. d/b/a TrueBlue Clinical Research, Tampa, Florida
  - Care Access - Tampa, Tampa, Florida
  - American Clinical Trials - Acworth, Acworth, Georgia
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Emory University School of Medicine, Atlanta, Georgia
  - Fides Clinical Research, Atlanta, Georgia
  - Southeastern Clinical Research Institute, Augusta, Georgia
  - American Clinical Trials - Douglasville, Douglasville, Georgia
  - Center for Advanced Research & Education, Gainesville, Georgia
  - The Jones Center Clinical Research, Macon, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - Clinical Investigation Specialists, Gurnee, Illinois
  - Nephrology Associates of Northern Illinois and Indiana (NANI) - Hinsdale, Hinsdale, Illinois
  - Accellacare - DuPage, Lombard, Illinois
  - Alliance for Multispecialty Research, LLC, Park Ridge, Illinois
  - Rockford Nephrology Associates, Rockford, Illinois
  - Central Illinois Diabetes and Clinical Research a Division of Prairie Education and Research Cooperative, Springfield, Illinois
  - Qualmedica Research, LLC, Evansville, Indiana
  - Nephrology Associates of Northern Illinois and Indiana (NANI) - Fort Wayne, Fort Wayne, Indiana
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Nephrology Associates of Northern Illinois and Indiana - IKS - Indianapolis South, Indianapolis, Indiana
  - Care Access - South Indianapolis, Indianapolis, Indiana
  - Reid Physician Associates, Richmond, Indiana
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - The University of Kansas - Clinical Research Center, Fairway, Kansas
  - Alliance for Multispecialty Research, LLC, Newton, Kansas
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Cotton O'Neil Diabetes & Endocrinology, Topeka, Kansas
  - Qualmedica Research, Bowling Green, Kentucky
  - Alliance for Multispecialty Research, LLC, Lexington, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - Care Access - Lake Charles, Lake Charles, Louisiana
  - IMA Clinical Research Monroe - Armand, Monroe, Louisiana
  - Alliance for Multispecialty Research, LLC, New Orleans, Louisiana
  - Sinai Hospital Of Baltimore, Baltimore, Maryland
  - Care Access - Baltimore, Baltimore, Maryland
  - Ascension Saint Agnes Heart Care, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - Jadestone Clinical Research, Beltsville, Maryland
  - Anderson Medical Research, Ft. Washington, Maryland
  - MedStar Health Research Institute (MedStar Physician Based Research Network), Hyattsville, Maryland
  - NECCR PrimaCare Research, Fall River, Massachusetts
  - Care Access - Quincy, Quincy, Massachusetts
  - Revival Research Institute, LLC, Dearborn, Michigan
  - Elixia MKC, LLC, Pontiac, Michigan
  - Lake Michigan Nephrology, Saint Joseph, Michigan
  - Great Lakes Research Institute, Southfield, Michigan
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Alliance for Multispecialty Research, LLC, Kansas City, Missouri
  - Clinvest Headlands Llc, Springfield, Missouri
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Boeson Research MSO, Missoula, Montana
  - Henderson Clinical Trials, Henderson, Nevada
  - DaVita Clinical Research - Las Vegas, Las Vegas, Nevada
  - Excel Clinical Research, LLC, Las Vegas, Nevada
  - Alliance for Multispecialty Research, LLC, Las Vegas, Nevada
  - Advanced Biomedical Research of America - South Eastern Avenue, Las Vegas, Nevada
  - Vector Clinical Trials, Las Vegas, Nevada
  - Albany Medical College, Division of Community Endocrinology, Albany, New York
  - Capital Cardiology Associates, Albany, New York
  - Westchester Medical Center Advanced Physicians Service, Kingston, New York
  - St. Francis Hospital & Heart Center, New Hyde Park, New York
  - NYU Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Saratoga Clinical Research, Saratoga Springs, New York
  - Care Access - Fayetteville, Fayetteville, North Carolina
  - Medication Management, Greensboro, North Carolina
  - Physician's East Endocrinology, Greenville, North Carolina
  - IMA Clinical Research - Lenoir, Lenoir, North Carolina
  - West Clinical Research, Morehead City, North Carolina
  - Accellacare - Raleigh, Raleigh, North Carolina
  - Accellacare - Wilmington - 1917 Tradd Court, Wilmington, North Carolina
  - Advanced Medical Research, Maumee, Ohio
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - Heritage Valley Multispecialty Group, Inc, Beaver, Pennsylvania
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Clinical Renal Associates Ltd., Media, Pennsylvania
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - Tristar Clinical Investigations, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Preferred Clinical Research-St. Clair, Pittsburgh, Pennsylvania
  - Guthrie Medical Group, P.C., Sayre, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Walker Family Care, Little River, South Carolina
  - Care Access - Mauldin, Mauldin, South Carolina
  - Circle Clinical Research, Sioux Falls, South Dakota
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Care Access - Memphis 2, Memphis, Tennessee
  - IMA Clinical Research Austin, Austin, Texas
  - Headlands Research - Brownsville, Brownsville, Texas
  - South Texas Clinical Research, Corpus Christi, Texas
  - Private Practice - Dr. Osvaldo A. Brusco, Corpus Christi, Texas
  - Baylor Soltero CV Research Center, Dallas, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Renal Disease Research Institute, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Soma Clinical Trials, Denison, Texas
  - South Texas Research Institute, Edinburg, Texas
  - Medresearch Inc, El Paso, Texas
  - Diabetes and Thyroid Center of Ft. Worth, Fort Worth, Texas
  - Valley Institute of Research - Fort Worth, Fort Worth, Texas
  - Juno Research, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Aqua Research Institute, Houston, Texas
  - Northwest Houston Cardiology - Cypress, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Research Physicians Network, LLC, Houston, Texas
  - Accurate Clinical Research, Inc, Humble, Texas
  - Texas Institute for Kidney and Endocrine Disorders, Lufkin, Texas
  - Wellness Clinical Research, McKinney, Texas
  - Revival Research Institute, LLC, McKinney, Texas
  - PRX Research, Mesquite, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Clinical Advancement Center, San Antonio, Texas
  - Discovery Clinical Trials - San Antonio, San Antonio, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - DaVita Clinical Research - North Houston, Shenandoah, Texas
  - Medrasa Clinical Research, Wylie, Texas
  - Alpine Research Organization, Clinton, Utah
  - Alliance for Multispecialty Research, LLC, Layton, Utah
  - Synexus Clinical Research US, Inc., Salt Lake City, Utah
  - Utah Kidney Research Institute, Salt Lake City, Utah
  - Alliance for Multispecialty Research, LLC, Norfolk, Virginia
  - Dominion Medical Associates, Inc., Richmond, Virginia
  - Eastside Research Associates, Redmond, Washington
  - Universal Research Group, Tacoma, Washington
  - IMA Clinical Research West Virginia, Morgantown, West Virginia
  - St. Vincent Hospital d/b/a Prevea Health, Green Bay, Wisconsin
  - Clinical Investigation Specialists, Kenosha, Wisconsin
- Argentina (58):
  - CONEXA Investigacion Clinica S.A., Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - Buenos Aires Macula S.A, Buenos Aires
  - Consultorio de Investigación Clínica EMO SRL, Buenos Aires
  - Cardiología Palermo, Buenos Aires
  - Stat Research S.A., Buenos Aires
  - Investigaciones Medicas Imoba Srl, Buenos Aires
  - CIPREC, Buenos Aires
  - Centro Médico Viamonte, Buenos Aires
  - Mautalen Salud e Investigación, Buenos Aires
  - CEMEDIC, Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires
  - Fundación Respirar, Buenos Aires
  - Glenny Corp. S.A., Buenos Aires
  - CEMEDIAB, C.a.b.a.
  - CEDIC, CABA
  - Instituto Médico Especializado (IME), CABA
  - Centro Medico Privado CEMAIC, Capital
  - IDIM - Instituto de Investigaciones Metabólicas, Ciudad de Buenos Aires
  - Centro Diabetológico Dr. Waitman, Córdoba
  - Instituto de Investigaciones Clínicas Córdoba, Córdoba
  - Sanatorio Privado Duarte Quirós, Córdoba
  - Centro Médico Colón, Córdoba
  - Centro Medico Privado San Vicente Diabetes, Córdoba
  - CIDIM-Centro Integral de Diagnostico por Imagenes Marchegiani, Córdoba
  - CIPADI - Centro Integral de Prevencion y Atencion en Diabetes, Godoy Cruz
  - Centro de Investigaciones Clínicas Baigorria, Granadero Baigorria
  - CMD-Centro Médico y Diagnóstico por Imágenes, Junín
  - Hospital Italiano de La Plata, La Plata
  - CIMeL, Lanús
  - Polo de Salud Vistalba, Luján de Cuyo
  - Centro de Investigaciones Médicas Mar del Plata, Mar del Plata
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata
  - Instituto De Investigaciones Clinicas Quilmes, Quilmes
  - DIM Clínica Privada, Ramos Mejía
  - Instituto Médico Río Cuarto, Río Cuarto
  - Fundacion Estudios Clinicos, Rosario
  - INECO Neurociencias Oroño, Rosario
  - Instituto Especialidades de la Salud Rosario, Rosario
  - Instituto Médico Catamarca IMEC, Rosario
  - Instituto Médico Fundación Grupo Colaborativo Rosario Investigación y Prevención Medica, Rosario
  - Instituto de Investigaciones Clinicas Rosario, Rosario
  - Laboratorio de Hemostasia y Trombosis, Rosario
  - Hospital Provincial del Centenario, Rosario
  - Centro de Investigaciones Médicas Tucuman, SAN M. de Tucuman
  - Corporación Médica San Martín, San Martín
  - Centro Modelo de Cardiología, San Miguel de Tucumán
  - Investigaciones Clínicas Tucumán, San Miguel de Tucumán
  - Go Centro Medico San Nicolás, San Nicolás
  - Centro de Diagnóstico y Rehabilitación (CEDIR), Santa Fe
  - Clínica de Nefrología, Urología y Enfermedades Cardiovasculares, Santa Fe
  - Centro de Investigaciones Clinicas del Litoral, Santa Fe
  - Centro de Salud e Investigaciones Médicas, Santa Rosa
  - Sanatorio Norte, Santiago del Estero
  - Centro de Investigaciones Medicas Temperley, Temperley
  - Sanatorio San Martin, Venado Tuerto
  - CEREHA, Villa Domínico
  - Instituto de Investigaciones Clinicas Zarate, Zárate
- Australia (16):
  - Nightingale Research, Adelaide
  - Emeritus Research, Botany
  - Box Hill Hospital, Box Hill
  - Royal Brisbane and Women's Hospital, Brisbane
  - Northern Beaches Clinical Research, Brookvale
  - Emeritus Research, Camberwell
  - Canberra Hospital, Garran
  - Barwon Health, Geelong
  - Austin Health - Repatriation Hospital, Heidelberg West
  - Logan Hospital, Meadowbrook
  - The Alfred Hospital, Melbourne
  - The AIM Centre / Hunter Diabetes Centre, Merewether
  - Fiona Stanley Hospital, Murdoch
  - Southern Adelaide Diabetes & Endocrine Services, Oaklands Park
  - Royal North Shore Hospital, St Leonards
  - University of Sydney - Charles Perkins Centre, Sydney
- Austria (12):
  - Krankenhaus St. Josef Braunau, Braunau am Inn
  - VIVIT, Feldkirch
  - Medizinische Universität Graz, Graz
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Konventhospital der Barmherzigen Brüder Linz, Linz
  - Cardio Metabolic Centre, Mattersburg
  - Private Practice - Dr. Evelyn Fliesser-Gorzer, Sankt Stefan ob Stainz
  - Klinik Landstraße, Vienna
  - Zentrum für klinische Studien Dr Hanusch Gmbh, Vienna
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
  - Klinik Hietzing, Vienna
  - Imed19-privat, Vienna
- Belgium (21):
  - AZORG Campus Aalst-Moorselbaan, Aalst
  - ANIMA Research, Alken
  - Imelda General Hospital, Bonheiden
  - Algemeen Ziekenhuis klina, Brasschaat
  - Centre Hospitalier Universitaire Brugmann, Brussels
  - Université Libre de Bruxelles - Hôpital Erasme, Brussels
  - UZ Brussel, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - Antwerp University Hospital, Edegem
  - UZ Gent, Ghent
  - Jessa Ziekenhuis, Hasselt
  - Jan Yperman Ziekenhuis, Ieper
  - Kormont, Kluisbergen
  - AZ Groeninge Campus Kennedylaan, Kortrijk
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman, Liège
  - ZNA Jan Palfijn, Merksem
  - Az Damiaan vzw, Ostend
  - Artsenpraktijk OHIO, Oudenaarde
  - Private Practice - Dr. De Watertoren, Tielt
  - Private Practice - Dr. Tim Decraecke (Zwalm), Zwalm
- Brazil (48):
  - Centro de Pesquisa Clinica do Coracao, Aracaju
  - Hospital Universitário João de Barros Barreto, Belém
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - Freire Pesquisa Clínica, Belo Horizonte
  - AngioKormann Blumenau, Blumenau
  - L2IP - Instituto de Pesquisas Clínicas, Brasília
  - Chronos Pesquisa Clínica, Brasília
  - Instituto de Pesquisa clinica de Campinas, Campinas
  - Centro de Pesquisa Sao Lucas, Campinas
  - Centro de Endocrinologia Geloneze, Campinas
  - Fundação Universidade de Caxias do Sul (FUCS), Caxias do Sul
  - Cline Research Center, Curitiba
  - Quanta Diagnóstico e Terapia, Curitiba
  - PUC Trials- Nucleo de Pesquisa clinica da Escola de Medicina da PUCPR, Curitiba
  - Instituto Pro Renal Brasil, Curitiba
  - Centro de Diabetes Curitiba, Curitiba
  - Instituto de Ensino e Pesquisa Clinica do Ceara, Fortaleza
  - Instituto de Estudos e Pesquisas Clinicas do Ceara IEP-CE, Fortaleza
  - Private Practice - Dr.Miguel N. Hissa, Fortaleza
  - Universidade Federal de Goias, Goiânia
  - Centro de Pesquisas Clínicas Dr. Marco Mota, Maceió
  - CPHOSP Manaus Medicina, Ensino e Pesquisa, Manaus
  - Centro de Pesquisa Clínica de Marília - CPCLIM, Marília
  - Instituto Méderi de Pesquisa e Saúde, Passo Fundo
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul, Porto Alegre
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - Ruschel Medicina e Pesquisa Clínica, Rio de Janeiro
  - Hospital Pro-Cardiaco, Rio de Janeiro
  - Clinica Senhor do Bonfim CSB - Salvador, Salvador
  - Pesquisare Saude, Santo André
  - Praxis Pesquisa Medica, Santo André
  - Centro Multidisciplinar de Estudos Clinicos, São Bernardo do Campo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
  - ISPEM - Instituto São José dos Campos em Pesquisas Médicas, São José dos Campos
  - Instituto de Pesquisa Clinica, São Paulo
  - CPQuali Pesquisa Clínica, São Paulo
  - CPCLIN, São Paulo
  - BR Trials - Ensaios Clinicos e Consultoria, São Paulo
  - BP - A Beneficencia Portuguesa de São Paulo, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - IBCC - Núcleo de Pesquisa e Ensino, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
  - Hospital das Clinicas FMUSP, São Paulo
  - Incor - Instituto do Coracao, São Paulo
  - Instituto de Molestias Cardiovasculares de Tatui, Tatuí
  - Eurolatino Pesquisas Medicas, Uberlândia
  - CEDOES, Vitória
  - Integral Pesquisa e Ensino, Votuporanga
- Canada (22):
  - C-health Research, Calgary
  - Ecogene-21, Chicoutimi
  - Med Trust Research, Courtice
  - C-health, Edmonton
  - St. Joseph's Health Care, London
  - Victoria Hospital & Children's Hospital - London Health Sciences Centre, London
  - Western Centre for Public Health and Family Medicine, London
  - G A Research Associates, Moncton
  - North York Diagnostic and Cardiac Centre, North York
  - Lakeridge Health, Oshawa
  - Alpha Recherche Clinique, Québec
  - Unité de Recherche Clinique du CISSS des Laurentides, Saint-Jérôme
  - Ocean West Research Clinic, Surrey
  - SMH Cardiology Clinical Trials, Surrey
  - Care Access - Cape Breton, Sydney
  - Care Access - Thunder Bay - Barton Street, Thunder Bay
  - Corcare, Toronto
  - Toronto General Hospital, Toronto
  - Clinical Research Solutions - Kitchener, Waterloo
  - Winchester District Memorial Hospital, Winchester
  - Seven Oaks General Hospital, Winnipeg
  - Winnipeg Clinic, Winnipeg
- Czechia (31):
  - MEDICUS SERVICES s.r.o., kardiologicka ambulance, Brandýs nad Labem
  - Fakultni Nemocnice u sv. Anny v Brne, Brno
  - UNIVMED, Brno
  - Vojenská Nemocnice Brno, Brno
  - Kardio Chlumec, Chlumec nad Cidlinou
  - Nemocnice Cesky Krumlov, Český Krumlov
  - Diahaza s.r.o., Holešov
  - Kardioma, Kolín
  - Kardiologicka ambulance, Litovel
  - EDUMED - Náchod, Náchod
  - Agentura Science Pro, Olomouc
  - Diabetologicke centrum s.r.o., Olomouc
  - PreventaMed, Olomouc
  - Private Practice - Dr. Miroslav Koliba, Ostrava
  - VASOMED Clinic, Ostrava
  - Kardiologicka a Angiologicka Ambulance, Ostrava - Dubina
  - MUDr. Jana Parkanyiova, Prague
  - Synexus Czech, Prague
  - MEDICON, Prague
  - Fakultni Thomayerova nemocnice, Prague
  - Nefrologie, Prague
  - Poliklinika Lípa Centrum, Prague
  - FLEDIP - Na dlouhem lanu, Prague
  - Centrum Kardiovaskularni Mediciny, Prague
  - Diabetologie a endokrinologie, J.Venerová, Prague
  - ResTrial s.r.o., Prague
  - MUDr. Barbora Diepoltova, Praha 9 - Klanovice
  - Diakom, s.r.o. - Přeštice, Přeštice
  - Kardiologicka ambulance MUDr. Ferkl s.r.o., Trutnov
  - Clinical Trials Service s.r.o., Uherské Hradiště
  - Cardio Research, s.r.o, Zlín
- Denmark (6):
  - Sygehus Sønderjylland i Aabenraa, Aabenraa
  - Aarhus Universitetshospital, Skejby, Aarhus
  - Sanos Clinic - Nordjylland, Gandrup
  - Herlev and Gentofte Hospital, Herlev
  - Sanos Clinic, Herlev
  - Sanos Clinic - Syddanmark, Vejle
- France (16):
  - Centre Hospitalier Universitaire - Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Bois-Guillaume
  - Bordeaux University Hospital - Pellegrin, Bordeaux
  - Chu Gabriel Montpied, Clermont-Ferrand
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Chu Grenoble Alpes, La Tronche
  - Centre Hospitalier Louis Pasteur, Le Coudray
  - CHU Montpellier Lapeyronie Hospital, Montpellier
  - Hôpital Nord Guillaume-et-René-Laennec / CHU de Nantes, Nantes
  - Centre Hospitalier Universitaire de Nice - Hopital Pasteur, Nice
  - Pitie Salpetriere University Hospital, Paris
  - Groupe hospitalier Paris saint Joseph, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - CHU Bordeaux Haut-Leveque, Pessac
  - CHU Rangueil, Toulouse
  - Centre Hospitalier Régional Universitaire de Tours - Hôpital Bretonneau, Tours
  - Polyclinique Vauban, Valenciennes
- Germany (25):
  - Kerckhoff-Klinik, Bad Nauheim
  - Herz - und Diabeteszentrum Nordrhein - Westfalen, Bad Oeynhausen, Bad Oeynhausen
  - FutureMeds GmbH, Berlin
  - Kardiologisch-Angiologische Praxis - Herzzentrum Bremen, Bremen
  - St.-Johannes-Hospital Dortmund, Dortmund
  - Hausärztlich-Kardiologisches MVZ am Felsenkeller GmbH/Zentrum für klinische Studien, Dresden
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - ZKS Suedbrandenburg, Elsterwerda
  - InnoDiab Forschung Gmbh, Essen
  - Unterfrintroper Hausarztzentrum Klinische Forschung, Essen
  - Universitätsklinikum Frankfurt Goethe-Universität, Frankfurt
  - Diabetes Zentrum Wilhelmsburg, Hamburg
  - Diabetes Zentrum Wandsbek, Hamburg
  - Zentrum für Nieren-, Hochdruck- und Stoffwechselerkrankungen - Heidering, Hanover
  - AmBeNet GmbH, Leipzig
  - Universität zu Lübeck - Institut für Endokrinologie und Diabetes, Lübeck
  - Universitätsmedizin Johannes Gutenberg Universität Mainz, Mainz
  - CRS Clinical Research Services Mannheim, Mannheim
  - Universitätsmedizin Mannheim, Mannheim
  - Institut für Diabetesforschung GmbH Münster, Münster
  - RED-Institut GmbH, Oldenburg
  - Kardiologische Praxis Papenburg, Papenburg
  - Zentrum für klinische Studien, Saint Ingbert
  - Nephrologisches Zentrum Villingen-Schwenningen, Villingen-Schwenningen
  - Praxis Sauter & Sauter & Vorbach, Wangen
- Greece (11):
  - Athens Medical Center - Psychikon branch, Athens
  - General Hospital of Athens "G. Gennimatas", Athens
  - General Hospital of Athens Laiko, Athens
  - Athens Medical Center, Athens
  - University Hospital of Ioannina, Ioannina
  - University General Hospital of Larissa, Larissa
  - Iatriko Paleou Falirou Medical Center, Palaió Fáliro
  - G. Gennimatas General Hospital of Thessaloniki, Thessaloniki
  - Euromedica General Clinic of Thessaloniki, Thessaloniki
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
  - 424 Military General Training Hospital, Thessaloniki
- Hungary (14):
  - DRC Gyógyszervizsgáló Központ, Balatongyörök
  - Szent Margit Rendelintézet, Budapest
  - Óbudai Egészségügyi Centrum, Budapest
  - Eszak-Pesti Centrumkorhaz-Honvedkorhaz, Budapest
  - PVN Kutató Kft, Budapest
  - Semmelweis University, Budapest
  - Privát Doktor Egészségügyi Zrt, Budapest
  - Újpesti Egészségügyi Nonprofit Kft, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - CRU Early Phase Unit, Kistarcsa
  - Selye János Kórház, Komárom
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged
  - Allergo-Derm Bakos Kft, Szolnok
  - Zala Megyei Szent Rafael Kórház, Zalaegerszeg
- India (19):
  - Motilal Nehru Medical College Hospital, Allahabād
  - Life Care Hospital and Research Centre, Bangalore
  - All India Institute of Medical Sciences, Bhubaneswar
  - Sardar Patel Medical College, Bikaner
  - Medway Hospitals - Kodambakkam, Chennai
  - Shri Mahant Indiresh Hospital, Dehradun
  - Endolife Speciality Hospitals, Guntur
  - K care Hospital, Kanpur
  - LPS Institute of Cardiology, Kanpur
  - Government Medical College - Kozhikode, Kozhikode
  - Dr. Ram Manohar Lohia Institute of Medical Sciences, Lucknow
  - Manipal Hospitals, Mysore
  - Kingsway Hospitals (Best Multispeciality Hospital in Nagpur), Nagpur
  - Shrikrishna Hrudayalaya And Critical Care Center, Nagpur
  - All India Institute of Medical Sciences (AIIMS) - Nagpur, Nagpur
  - G.B. Pant Institute of Postgraduate Medical Education & Research, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - Nirmal Hospital Pvt Ltd., Surat
  - Shri Bachubhai Dahyabhai Mehta Mahavir Heart Institute, Surat
- Israel (15):
  - Barzilai Medical Center, Ashkelon
  - Rambam Health Care Campus, Haifa
  - Bnai Zion Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
  - Rabin Medical Center - Hasharon Campus, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Sourasky Medical Center, Tel Aviv
  - Maccabi Healthcare Services, Tel Aviv
  - Diabetes Medical Center, Tel Aviv
  - Yitzhak Shamir Medical Center, Ẕerifin
- Italy (14):
  - IRCCS - AOU di Bologna, Bologna
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna
  - Azienda Ospedaliero Universitaria S.Anna, Ferrara
  - Ospedale San Martino, Genova
  - Centro Cardiologico Monzino, Milan
  - Ospedale San Raffaele, Milan
  - A.O.U. Policlinico Paolo Giaccone, Palermo
  - AO Santa Maria della Misericordia, Perugia
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - AOU Policlinico Umberto I, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Roma
  - Fondazione Policlinico Universitario Campus Bio-Medico, Rome
  - IRCCS Policlinico San Donato, San Donato Milanese
- Mexico (42):
  - Centro de Atencion al Diabetico Actopan, Actopan
  - Fundación Cardiovascular de Aguascalientes A.C., Aguascalientes
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, Ciudad Madero
  - Cryptex Investigación Clínica S.A. de C.V., Cuauhtémoc, Ciudad de México
  - Instituto de Diabetes, Obesidad y Nutricion, Cuernavaca
  - Investigación Clínica Cuernavaca, S.C., Cuernavaca
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Lahoja. Asociacion Para La Investigacion Y La Farmacovigilancia, Durango
  - Instituto Jalisciense de Investigacion en Diabetes y Obesidad, Guadalajara
  - Diseno y Planeacion en Investigacion Medica, Guadalajara
  - Centro de Investigación Clínica y Medicina Traslacional (CIMeT), Guadalajara
  - Private Practice - Dr. Arechavaleta Granell Maria del Rosario, Guadalajara
  - Virgen Cardiovascular Research SC, Guadalajara
  - CINVEC Medica, Guadalajara
  - Instituto Cardiovascular de León S.C., León
  - Centro de Investigacion en Artritis y Osteoporosis SC, Mexicali
  - Clínicos Asociados BOCM, Mexico City
  - Hospital de Jésus, I.A.P., Mexico City
  - Clinica Omega, Mexico City
  - Centro Especializado En Diabetes, Obesidad Y Prevencion De Enfermedades Cardiovasculares, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - EME RED Hospitalaria, Mérida
  - Medical Care and Research SA de CV, Mérida
  - Clinstile, S.A. de C.V., México
  - Instituto Nacional de Cardiologia Ignacio Chavez, México
  - Servicios de Oncología Medica Integral - Monterrey - José Benitez, Monterrey
  - Cardiolink Clin Trials, Monterrey
  - IMED Internal Medicine Clin Trials, Monterrey
  - UBAM Unidad Biomedica Avanzada Monterrey, Monterrey
  - Clínica García Flores SC, Monterrey
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City
  - Boca Clinical Trials Mexico SC, Puebla City
  - Centro de Estudios Clínicos de Querétaro (CECLIQ), Querétaro
  - PanAmerican Clinical Research - Querétaro - Avenida Antea, Querétaro
  - Centro de Atención e Investigación Cardiovascular del Potosí, San Luis Potosí City
  - Centro de investigación y control metabólico, San Nicolás de los Garza
  - Medimanage Research, Tlalpan
  - Instituto Veracruzano en Investigación Clínica S.C., Veracruz
  - Arké SMO S.A de C.V, Veracruz
  - FAICIC S. de R.L. de C.V., Veracruz
  - Consultorio de Medicina Especilizada del Sector Privado, Xalapa
- Netherlands (28):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - EB Medical Research, Almere Stad
  - Meander Medisch Centrum, Amersfoort
  - OLVG Oost, Amsterdam
  - Amsterdam UMC, locatie AMC, Amsterdam
  - Gelre Ziekenhuis, Apeldoorn
  - Rode Kruis Ziekenhuis, Beverwijk
  - Amphia Ziekenhuis, locatie Breda Molengracht, Breda
  - Het Van Weel-Bethesda Ziekenhuis - Ziekenhuis Dirksland, Dirksland
  - Albert Schweitzer Ziekenhuis, locatie Dordwijk, Dordrecht
  - Ziekenhuis Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Spaarne Gasthuis, Haarlem Zuid, Haarlem
  - Atrium-Orbis - Zuyderland Medisch Centrum Heerlen, Heerlen
  - Ziekenhuis Bethesda, Hoogeveen
  - Medische Centrum Leeuwarden, Leeuwarden
  - Radboudumc, Nijmegen
  - Bravis Ziekenhuis, locatie Roosendaal, Roosendaal
  - Franciscus Gasthuis & Vlietland, Locatie Gasthuis, Rotterdam
  - Medisch Centrum Thomsonplein, The Hague
  - Huisartsenpraktijk Disha, The Hague
  - Ziekenhuis Rivierenland, Tiel
  - Universitair Medisch Centrum Utrecht, Utrecht
  - VieCuri Medisch Centrum, locatie Venlo, Venlo
  - Huisartsenpraktijk Broekman, Zwijndrecht
  - Dokters van Nederhoven, Zwijndrecht
  - Isala, locatie Zwolle, Zwolle
- New Zealand (8):
  - Pacific Clinical Research Network - Auckland (PCRN Auckland), Auckland
  - Aotearoa Clinical Trials, Auckland
  - Pacific Clinical Research Network - Tasman, Nelson
  - Lakeland Clinical Trials Culloden, Papamoa
  - Momentum Clinical Research - Pukekohe, Pukekohe
  - PCRN Silverdale Medical, Silverdale
  - Lakeland Clinical Trials Wellington, Upper Hutt
  - Aotearoa Clinical Trials - Whangarei, Whangarei
- Poland (20):
  - KLIMED Marek Klimkiewicz, Bialystok
  - Polsko-Amerykańskie Kliniki Serca II Oddział Kardiologiczny, Bielsko-Biala
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - Centrum Medyczne INTERCOR Sp. z o.o., Bydgoszcz
  - Diab Serwis Popenda Spółka Jawna, Chorzów
  - Polsko-Amerykańskie Kliniki Serca PAKS Małopolskie Centrum Sercowo-Naczyniowe, Chrzanów
  - Centrum Kliniczno-Badawcze, Elblag
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Medyczne Centrum Diabetologiczno Endokrynologiczno Metaboliczne DIAB-ENDO-MET, Krakow
  - Poliklinika Kardiologiczna Serce, Leszno
  - Pro Salus Centrum Medyczne, Lodz
  - CenterMed Lublin NZOZ, Lublin
  - Ekamed, Lublin
  - EndoPractica, Opole
  - Centrum Zdrowia Metabolicznego Pawel Bogdanski, Poznan
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu, Przemyśl
  - Centrum Szybkiej Diagnostyki Kardiologicznej "Kardiomed" M. Żabówka E. Żabówka, Tarnów
  - Polsko-Amerykańskie Kliniki Serca, Tychy
  - Balsam Medica, Warsaw
  - NZOZ Centurm Medyczne SERAFIN-MED, Żarów
- Puerto Rico (3):
  - Advanced Clinical Research, LLC, Bayamón
  - Clinical Research Management Group Inc, Ponce
  - GCM Medical Group, PSC - Hato Rey Site, San Juan
- Romania (21):
  - Private Practice - Dr. Mercea Corina Delia, Baia Mare
  - CMI DNBM Dr. Pop Lavinia, Baia Mare
  - C.M.D.T.A. Neomed, Brasov
  - Nicodiab, Bucharest
  - Hightech Medical Services SRL-Centrul pentru Studiul Metabolismului, Bucharest
  - Centrul Medical NutriLife, Bucharest
  - Lotus-Med Tunari, Bucharest
  - Centrul Medical Endocrinologie si Diabet Dr. Paveliu, Bucharest
  - Spitalul Clinic Județean de Urgență, Craiova
  - Milena Sante, Galați
  - Diamed Obesity, Galați
  - Centrul Medical Consultmed, Iași
  - Cardiomed Iași, Iași
  - Clinica Korall, Satu Mare
  - Policlinica Astra Sibiu, Sibiu
  - SC Dentosim Queen SRL - Centrul Medical Diamed, Târgu Mureş
  - Centrul Medical Mediab, Târgu Mureş
  - Mediab S.R.L., Târgu Mureş
  - Cabinet Medical Dr.Geru, Timișoara
  - Institutul de Boli Cardiovasculare Timișoara, Timișoara
  - Centrul Medical Medicalis, Timișoara
- Slovakia (18):
  - Cliniq s.r.o., Bratislava
  - ENDIAMED s.r.o, Dolný Kubín
  - JM-Interna s.r.o, Dolný Kubín
  - IN-DIA, Lučenec
  - Nemocnica s poliklinikou Lucenec, Lučenec
  - NEDÚ - Národný endokrinologický a diabetologický ústav n.o., Ľubochňa
  - Sin Azucar, Malacky
  - AMBORA s.r.o. Interna ambulancia, Martin
  - B-Medical, s.r.o., Námestovo
  - Fakultná nemocnica Nitra, Nitra
  - FUNKYSTUFF s.r.o., Nové Zámky
  - MEDIKALS, Piešťany
  - MUDr. Judita Gondova, Poltár
  - ENRIN, s.r.o., Rimavská Sobota
  - Tatratrial s.r.o., Rožňava
  - Areteus s.r.o., Trebišov
  - MediPrax, s.r.o., Trstená
  - IRIDIA, Vrútky
- Spain (14):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña
  - Centro Periférico de Especialidades Bola Azul, Almería
  - Hospital Universitario de La Ribera, Alzira
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Complejo Hospitalario Universitario de Ferrol (CHUF)- Hospital Naval, Ferrol
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Clínica Juaneda, Palma de Mallorca
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Clínica nuevas Tecnologías en Diabetes y Endocrinología (NTDE), Seville
  - Hospital Quiron Infanta Luisa, Seville
  - Vithas Hospital Sevilla, Seville
  - Hospital Universitario Doctor Peset, Valencia
- Turkey (Türkiye) (21):
  - Afyon Kocatepe Üniversitesi Tıp Fakültesi, Afyonkarahisar
  - Ankara Bilkent Şehir Hastanesi, Ankara
  - Hacettepe Universite Hastaneleri, Ankara
  - Akdeniz Universitesi Hastanesi, Antalya
  - Ege Universitesi Hastanesi, Bornova
  - T.C. Saglik Bakanligi - Hitit Universitesi Corum Egitim ve Arastirma Hastanesi, Çorum
  - Trakya University Medical Faculty Hospital, Edirne
  - Eskisehir Osmangazi University, Eskişehir
  - Gaziantep Universitesi Sahinbey Arastirma ve Uygulama Hastanesi, Gaziantep
  - Dr. Siyami Ersek Göğüs Kalp Ve Damar Cerrahisi Eğitim Ve Araştırma Hastanesi, Istanbul
  - Kartal Koşuyolu Yüksek İhtisas Eğitim ve Araştirma Hastanesi, Istanbul
  - Istanbul Universitesi Cerrahpasa, Istanbul- Fatih
  - Kocaeli Üniversitesi, İzmit
  - Erciyes Universitesi Tıp Fakultesi Hastaneleri, Kayseri
  - Kocaeli Üniversitesi, Kocaeli
  - Necmettin Erbakan University Meram Medical Faculty, Konya
  - T.C. Saglik Bakanligi - Dumlupinar Universitesi Kutahya Evliya Celebi Egitim ve Arastirma Hastanesi, Kütahya
  - Mersin University, Mersin
  - Ondokuz Mayıs Universitesi, Samsun
  - Cumhuriyet Universitesi, Sivas
  - Bursa Yüksek İhtisas Eğitim Ve Araştırma Hastanesi, Yıldırım
- Ukraine (15):
  - Regional Communal Non-commercial enterprise "Chernivtsi regional clinical hospital", Chernivtsi
  - Vise Clinic, Ivano-Frankivsk
  - Clinical Diagnostic Center, Ivano-Frankivsk
  - Institute of Endocrinology and Metabolism named after Komissarenko, Kiev
  - Edelweiss Medics, Kyiv
  - Medbud Clinic, Kyiv
  - Medical Center "Universal Clinic "Oberig" of Limited Liability Company "Kapytal", Kyiv
  - ARTEM, Kyiv
  - Center of Family Medicine Plus, Kyiv
  - Lviv City Clinical Hospital #4, Lviv
  - Branch "Center of Endocrinological Health" of "Lviv Regional Clinical Diagnostic Center", Lviv
  - Medical center Pulse in Vinnitsi, Vinnytsia
  - Limited liability company "Medical center Health Clinic", Vinnytsia
  - Vinnytsia Regional Clinical Endocrinology Dispensary, Vinnytsia
  - Communal Enterprise "Hospital #1" of Zhytomyr City Council, Zhytomyr
- United Kingdom (18):
  - Aberdeen Royal Infirmary, Aberdeen
  - FutureMeds - Birmingham, Birmingham
  - FutureMeds - Liverpool, Bromborough
  - University Hospital Coventry & Warwickshire, Coventry
  - FutureMeds Glasgow - CPS Research, Glasgow
  - Hull Royal Infirmary, Hull
  - Ipswich Hospital, Ipswich
  - Ashton Medical Group - Chapel House, Lancashire
  - Royal London Hospital, London
  - Altnagelvin Area Hospital, Londonderry
  - Futuremeds-Newcastle, Newcastle
  - Newquay Health Centre, Newquay
  - Homecroft Surgery, Redruth
  - FutureMeds Teesside - Middlefield Centre, Stockton-on-Tees
  - Swansea University, Swansea
  - Musgrove Park Hospital, Taunton
  - Rame Group Practice, Torpoint
  - Moorgreen Hospital, West End

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Heerspink HJL, van Raalte DH, Bjornstad P, Bunck MC, Wu P, Tunali I, Milicevic Z, Koeneman L. Rationale, Design, and Baseline Characteristics of the TRANSCEND-CKD trial of Retatrutide in Patients with Chronic Kidney Disease. Nephrol Dial Transplant. 2025 Oct 29:gfaf230. doi: 10.1093/ndt/gfaf230. Online ahead of print. PMID 41160422
- See also: The Effect of Retatrutide Once Weekly on Cardiovascular Outcomes and Renal Function in Adults Living With Obesity (TRIUMPH-OUTCOMES) — https://trials.lilly.com/en-US/trial/479798